CLINICAL TRIAL: NCT03482661
Title: Magnetic Steering of Capsule Endoscopy Improves Small Bowel Capsule Endoscopy Completion Rate
Brief Title: Magnetic Steering Improves Small Bowel Capsule Endoscopy Completion Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuan Liao (Other)
Responsible Party: Sponsor-Investigator, Zhuan Liao, professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MCE-CECR
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Capsule Endoscopy; Small Bowel Disease
Keywords: Magnetic steering; MCE; CECR

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The patients swallowed the capsule with water in the supine position. When the capsule reached the stomach, the capsule was lifted away from the posterior wall, rotated and advanced to the fundus and cardiac regions, and then to the gastric body, angulus, antrum and pylorus. After completing the stomach examination, the capsule moved automatically without magnetic control and entered the duodenum under physiological conditions. The position of the capsule was verified through real-time viewer.
- Magnetic steering (Experimental): After finishing the stomach examination as the control protocol, the capsule was lifted with the magnetic control, then rotating the capsule until the camera end oriented toward the pylorus . Next, the endoscopist could drag the capsule close to the pylorus with the guidance magnet robot, waiting for the open of pylorus. Once the pylorus opened, the capsule could enter the duodenum with gastric peristalsis.
  Interventions: Other: magnetic steering

INTERVENTIONS:
Other: magnetic steering — The capsule was controlled to pass through the pylorus by magnet steering.
  Arms: Magnetic steering

SUMMARY:
Patients referred for magnetically controlled capsule endoscopy (MCE) in the participating center from June 2017 to November 2017 were prospectively enrolled. Magnetic steering of MCE was performed after standard gastric examination. Capsule endoscopy completion rate (CECR), gastric transit time (GTT), pyloric transit time (PTT) and rapid gastric transit rate (GTT ≤ 30 min) were compared with the historical control group enrolled from January 2017 to May 2017.

DETAILED DESCRIPTION:
Background and aims: Capsule endoscopy is currently available as a noninvasive and effective diagnostic modality to identify small bowel abnormalities, while the completion rate ranged from 75.1% to 95.6%. A novel magnetically controlled capsule endoscopy (MCE) system could facilitate the capsule to pass through pylorus thereby reducing the gastric transit time (GTT). The investigators perform this study to determine the potential improvement in capsule endoscopy completion rate (CECR) under magnetic steering vs standard mode.

Methods: Patients referred for magnetically controlled capsule endoscopy (MCE) in the participating center from June 2017 to November 2017 were prospectively enrolled. Magnetic steering of MCE was performed after standard gastric examination. Capsule endoscopy completion rate (CECR), gastric transit time (GTT), pyloric transit time (PTT) and rapid gastric transit rate (GTT ≤ 30 min) were compared with the historical control group enrolled from January 2017 to May 2017.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged over 18
* With gastrointestinal complaints
* Scheduled to undergo a capsule endoscopy for both stomach and small bowel

Exclusion Criteria:

* No surgical condition or refusing abdominal surgery to take out the capsule in case of capsule retention
* Implanted pacemaker, except the pacemaker is compatible with MRI
* Other implanted electromedical devices or magnetic metal foreign bodies
* Pregnancy or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
CECR | Two weeks
  Capsule endoscopy completion rate

SECONDARY OUTCOMES:
Diagnostic cases by MCE | Two weeks
  Esophageal, gastric, small bowel and colon diseases diagnosed by MCE
Transit time | Two weeks
  Esophageal/gastric/pyloric/small bowel/total transit time
Rapid gastric transit rate | Two weeks
  Rate of patients with a gastric transit time of ≤ 30 min

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
We may share IPD when we finish this research

REFERENCES:
- [Background] Tziatzios G, Gkolfakis P, Dimitriadis GD, Triantafyllou K. Long-term effects of video capsule endoscopy in the management of obscure gastrointestinal bleeding. Ann Transl Med. 2017 May;5(9):196. doi: 10.21037/atm.2017.03.80. PMID 28567376
- [Background] Kopylov U, Yung DE, Engel T, Vijayan S, Har-Noy O, Katz L, Oliva S, Avni T, Battat R, Eliakim R, Ben-Horin S, Koulaouzidis A. Diagnostic yield of capsule endoscopy versus magnetic resonance enterography and small bowel contrast ultrasound in the evaluation of small bowel Crohn's disease: Systematic review and meta-analysis. Dig Liver Dis. 2017 Aug;49(8):854-863. doi: 10.1016/j.dld.2017.04.013. Epub 2017 Apr 27. PMID 28512034
- [Background] Cheung DY, Kim JS, Shim KN, Choi MG; Korean Gut Image Study Group. The Usefulness of Capsule Endoscopy for Small Bowel Tumors. Clin Endosc. 2016 Jan;49(1):21-5. doi: 10.5946/ce.2016.49.1.21. Epub 2016 Jan 28. PMID 26855919
- [Background] Pennazio M, Spada C, Eliakim R, Keuchel M, May A, Mulder CJ, Rondonotti E, Adler SN, Albert J, Baltes P, Barbaro F, Cellier C, Charton JP, Delvaux M, Despott EJ, Domagk D, Klein A, McAlindon M, Rosa B, Rowse G, Sanders DS, Saurin JC, Sidhu R, Dumonceau JM, Hassan C, Gralnek IM. Small-bowel capsule endoscopy and device-assisted enteroscopy for diagnosis and treatment of small-bowel disorders: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2015 Apr;47(4):352-76. doi: 10.1055/s-0034-1391855. Epub 2015 Mar 31. PMID 25826168
- [Background] Liao Z, Gao R, Xu C, Li ZS. Indications and detection, completion, and retention rates of small-bowel capsule endoscopy: a systematic review. Gastrointest Endosc. 2010 Feb;71(2):280-6. doi: 10.1016/j.gie.2009.09.031. PMID 20152309
- [Background] Koulaouzidis A, Giannakou A, Yung DE, Dabos KJ, Plevris JN. Do prokinetics influence the completion rate in small-bowel capsule endoscopy? A systematic review and meta-analysis. Curr Med Res Opin. 2013 Sep;29(9):1171-85. doi: 10.1185/03007995.2013.818532. Epub 2013 Jul 11. PMID 23790243
- [Background] Prichard D, Ou G, Galorport C, Enns R. Sham Feeding with Bacon Does Not Alter Transit Time or Complete Examination Rate During Small Bowel Capsule Endoscopy. Dig Dis Sci. 2018 Feb;63(2):422-428. doi: 10.1007/s10620-017-4901-7. Epub 2018 Jan 4. PMID 29302875
- [Background] Ou G, Svarta S, Chan C, Galorport C, Qian H, Enns R. The effect of chewing gum on small-bowel transit time in capsule endoscopy: a prospective, randomized trial. Gastrointest Endosc. 2014 Apr;79(4):630-6. doi: 10.1016/j.gie.2013.08.038. Epub 2013 Oct 7. PMID 24112594
- [Background] Liao Z, Hou X, Lin-Hu EQ, Sheng JQ, Ge ZZ, Jiang B, Hou XH, Liu JY, Li Z, Huang QY, Zhao XJ, Li N, Gao YJ, Zhang Y, Zhou JQ, Wang XY, Liu J, Xie XP, Yang CM, Liu HL, Sun XT, Zou WB, Li ZS. Accuracy of Magnetically Controlled Capsule Endoscopy, Compared With Conventional Gastroscopy, in Detection of Gastric Diseases. Clin Gastroenterol Hepatol. 2016 Sep;14(9):1266-1273.e1. doi: 10.1016/j.cgh.2016.05.013. Epub 2016 May 20. PMID 27211503
- [Background] Zou WB, Hou XH, Xin L, Liu J, Bo LM, Yu GY, Liao Z, Li ZS. Magnetic-controlled capsule endoscopy vs. gastroscopy for gastric diseases: a two-center self-controlled comparative trial. Endoscopy. 2015 Jun;47(6):525-8. doi: 10.1055/s-0034-1391123. Epub 2015 Jan 15. PMID 25590177
- [Background] Zhu SG, Qian YY, Tang XY, Zhu QQ, Zhou W, Du H, An W, Su XJ, Zhao AJ, Ching HL, McAlindon ME, Li ZS, Liao Z. Gastric preparation for magnetically controlled capsule endoscopy: A prospective, randomized single-blinded controlled trial. Dig Liver Dis. 2018 Jan;50(1):42-47. doi: 10.1016/j.dld.2017.09.129. Epub 2017 Oct 6. PMID 29110963
- [Background] Albrecht H, Vetter M, Dauth W, Zoicas F, Neurath MF, Hagel AF. The impact of hospitalization on the performance of capsule endoscopy (CE). Dig Liver Dis. 2017 Jun;49(6):647-650. doi: 10.1016/j.dld.2017.02.010. Epub 2017 Feb 20. PMID 28258930
- [Derived] Luo YY, Pan J, Chen YZ, Jiang X, Zou WB, Qian YY, Zhou W, Liu X, Li ZS, Liao Z. Magnetic Steering of Capsule Endoscopy Improves Small Bowel Capsule Endoscopy Completion Rate. Dig Dis Sci. 2019 Jul;64(7):1908-1915. doi: 10.1007/s10620-019-5479-z. Epub 2019 Feb 6. PMID 30725289